CLINICAL TRIAL: NCT05997680
Title: A Parent-child Yoga Intervention for Reducing Attention Deficits in Children with Congenital Heart Disease: a Feasibility Study Prior to a Randomised Controlled Trial
Brief Title: A Parent-child Yoga Intervention for Reducing Attention Deficits in Children with Congenital Heart Disease: a Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Gallagher (Other)
Collaborators: Centre Universitaire de Santé McGill (Unknown); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor-Investigator, Anne Gallagher, Researcher and clinical neuropsychologist, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2020-2446; G-23-0033984 (Other Grant/Funding Number: Heart and Stroke Foundation of Canada)
Record Dates: First submitted 2023-08-02; First posted 2023-08-18 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Congenital Heart Disease; Child Development; Neurodevelopmental Disorders; Parents
Keywords: Neurodevelopment; Attention; Yoga; Motor Skills; Parenting Stress; Congenital Heart Disease
MeSH Terms: conditions — Heart Defects, Congenital; Neurodevelopmental Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The intervention team including the research coordinator will not be blinded to intervention allocation. The primary and secondary outcomes of the full trial will be assessed by a research assistant who is not part of the intervention and who will be blinded to intervention allocation. Data will be anonymised, and data quality control will be conducted by staff blinded to the intervention group. The intervention team will be blinded to the initial level of attention functioning. There will be no interference with standard clinical care. All clinical follow-up, therapies and learning-support services received as part of the standard clinical care will be documented in the electronic case report form. Due to the nature of the intervention, participants and their parents will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Yoga group (Experimental): Participants with CHD undergoing neurodevelopmental assessments and benefiting from the 8-week yoga intervention in addition to standard of care.
  Interventions: Behavioral: Parent-child yoga
- Waitlist control group (No Intervention): Participants with CHD undergoing neurodevelopmental assessments at the same time as the yoga group participants and benefiting from standard of care only during the 8 weeks of the intervention. The yoga intervention will be made available to all waitlist control group participants once their trial wave is completed.

INTERVENTIONS:
Behavioral: Parent-child yoga — The 45-minute yoga sessions are structured to include an opening and a closing ritual that remain the same throughout the 8 weeks, between which an active and a calming parts are scheduled. The active and calming parts are embedded in stories that align with the developmental level and interests typical of 4-to-6-year-olds. Each session is clearly structured with each exercise and transition well described in the Yoga for Little Hearts Yoga Program Manual. In addition to the yoga sessions, at-home exercises (5 min) including breathing, meditation and mindfulness activities will be explained to participants. We will ask them to practice them at home at least 3 times every week, for the 8-week duration of the intervention. Including the yoga session and home exercises, the 8-week intervention thus includes at least 60 minutes of yoga per week. Parents will be encouraged to pursue the at-home exercises after the end of the 8-week yoga program, up to the 6-month follow-up.
  Arms: Yoga group

SUMMARY:
The proposed study aims to determine the feasibility of the procedures for a future full randomized controlled trial (RCT), which will test the efficacy of a parent-child yoga intervention in reducing attention deficits in children with congenital heart disease (CHD). Specific aims of this single-blind, two-arm, two-center feasibility trial are to evaluate recruitment rates and capacity, withdrawal and dropout rates, adherence to the intervention, acceptability of the randomization process by families, variation in delivery of the intervention between yoga instructors, and standard deviation of main outcomes of the future RCT in order to determine its appropriate sample size. This feasibility study will lead to the first ever RCT to test the efficacy of an intervention strategy for reducing attention deficits in children with CHD. Ultimately, the implementation of this parent-child yoga program will lead to better long-term academic and psychosocial functioning and quality of life for these children and their family.

DETAILED DESCRIPTION:
Context

Congenital heart disease (CHD) is the most common structural birth defect, affecting up to 1% of newborns. Half of children with CHD present neurodevelopmental impairments, including significant attention deficits. Compared to the general population, they are at 2.5 to 4 times greater risk for attention deficit hyperactivity disorder (ADHD). Despite the high prevalence of these disabilities, very little interest has been given to the design and implementation of CHD-specific interventions for improving attention. In fact, only one randomised controlled trial (RCT) aimed at improving cognition in adolescents with CHD and revealed promising results for attention and inhibitory control. To date, no RCT aiming to improve attention has been conducted in young children with CHD, although attention has been strongly associated with school readiness and can predict academic skills. Yet, a rich literature supports the notion that early intervention is key to ensure success in the crucial first years of education. There is emerging evidence from RCTs indicating that parent-child yoga interventions improve attention and reduce ADHD symptoms in both typically developing and clinical populations. However, no studies have tested this promising approach in children with CHD although these children have their own challenges. Our ultimate goal is to test the efficacy of a parent-child yoga intervention to reduce attention deficits in children with CHD at school entry. Before launching a full RCT involving multiple sites across Canada, we propose to conduct the 2-site Yoga for Little Hearts feasibility study, which is a necessary and critical step to ensure future assessment and implementation of our parent-child yoga intervention program. Results from this feasibility study will allow us to optimize the subsequent large-scale RCT by preventing procedural and methodological issues.

Aims and hypotheses

The principal objectives of the proposed feasibility study are to evaluate: 1) recruitment rates and capacity; 2) retention, dropout and withdrawal rates during the 8-week parent-child yoga program and at 6-month follow-up; 3) adherence to the intervention; 4) acceptability of the randomisation process by families; 5) heterogeneity in the delivery of the intervention between yoga instructors, and use of home-based exercise between participants; 6) proportion of missing data in the standardized neurodevelopmental assessment instruments and parental questionnaires, and 7) standard deviation of primary outcomes of the full RCT in order to determine an appropriate sample size for the future full trial.

Following this feasibility study, we plan to conduct a full RCT including multiple centers aiming to test the efficacy of our 8-week parent-child yoga intervention in addition to the standard clinical care vs. standard clinical care alone in reducing attention deficits in 4-to-6-year-olds with CHD immediately and 6 months post-intervention.

Population

Children aged 4 to 6 years old with a diagnosis of CHD requiring heart surgery and their parents.

Procedure

The Yoga for Little Hearts feasibility methodology follows the Standard Protocol Items for Randomized Trials recommendations and the Consolidated Standards of Reporting Trials (CONSORT) statement - extension to randomized pilot and feasibility trials. Our proposed study is a single blind, two-center, two-arm randomized waitlist feasibility study. A total of 24 parent-child dyads, including children aged 4 to 6 years old with CHD, will be recruited in two centers and randomly assigned (2:1 allocation; 2 yoga intervention:1 standard of care) to receive either parent-child yoga intervention and standard clinical care (yoga intervention group) or standard clinical care alone with the opportunity to receive the yoga intervention after their participation in the study if desired (waitlist control group).

Two waves of recruitment of 6 parent-child dyads will be held in each of the two participating sites, for a total of 24 dyads recruited over an 18-month period. The two participating sites are the CHU Ste-Justine and the Montreal Children's Hospital (MCH), covering more than half of the pediatric population with CHD in the Québec province. For each recruitment wave and site, 4 of the 6 recruited dyads will receive an 8-week parent-child yoga intervention. Meanwhile, dyads allocated to the waitlist control group (2 of the 6 recruited dyads) will receive the standard of care only, with the opportunity to receive the yoga intervention when their participation in the study will be completed. All participants from the yoga intervention group (n = 16) and the waitlist control group (n = 8) will undergo 3 standardized interdisciplinary neurodevelopmental assessments: 1) at baseline, before randomization (T0); 2) immediately post-intervention (T1); 3) 6-month post-intervention (T2).

ELIGIBILITY:
To be eligible for the study, children need to meet the following inclusion criteria:

1. diagnosis of CHD requiring heart surgery;
2. aged 4 to 6 years old;
3. poor attentional skills measured with Variability score (0.5 standard deviation below norms) at the Kiddie Conners Continuous Performance Test, 2nd Edition (K-CPT2), a sensitive measure for attentional impairments. This inclusion criteria is important since yoga intervention has shown larger effects on attention in children with greater difficulties before the intervention;
4. parent willing to participate to the 8-week parent-child yoga intervention and the pre/post/6-month follow-up assessments;
5. for children with ADHD medication (approx. 5% of the 4-to-6-year-olds at our neurocardiac clinic), parent accept to temporary stop it to at least 48h prior to each assessment.

Exclusion criteria will be the following:

1. having a medical contraindication to the practice of yoga;
2. confirmed diagnosis of severe developmental or intellectual delay that would prevent successful completion of the planned study testing;
3. presence of severe physical handicap that would preclude the child from participating in the yoga intervention without special adaptation;
4. families who do not speak French or English (less than 3% of families followed in our clinics);
5. children who have been engaged in a structured weekly yoga program for at least a month in the past year (based on our parents' poll, less than 5%). However, parents included could have past or actual experience in practicing yoga.

Eligibility will be determined:

1. by consulting the child's medical record;
2. during a child medical visit at one of the sites or a virtual visit with the research team by administering the K-CPT2.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 2 months prior to the intervention.
  The number of eligible participants contacted, the number of consents to participation and the duration of the recruitment for each of the two waves of recruitment.
Dropout and withdrawal rates | The 8 weeks of the intervention.
  The number of eligible participants contacted, the number of consents to participation and the duration of the recruitment for each of the two waves of recruitment.
Adherence | The 8 weeks of the intervention.
  Adherence will be assessed by recording the number of sessions attended by each participant during the 8-week program. Acceptable adherence will be defined as completion of a minimum of 6/8 in-person yoga sessions otherwise the participant will be excluded from the analyses (withdrawals). Moreover, every week, parents will be asked to complete an at-home yoga exercise logbook to track the completion of yoga home practice and information will be collated at the end of the program.
Acceptability of the randomisation process | Months prior to the intervention.
  The number of refusals to enrol because of randomisation to intervention will be documented.
Variation in delivery of the intervention | The 8 weeks of the intervention.
  To document the variation between yoga instructors and sites, the instructors will complete an intervention logbook after each session checking all planned steps and exercises that have been completed and detailing all protocol deviations and their reasons. At the end of the 8-week program, the number of deviations, the moments and the groups in which they occurred, and their reasons will be documented in the feasibility form.
Missing data assessment | 2 weeks following each wave of assessments (T0, T1, T2).
  The missing data will be collected at the end of each neurodevelopmental assessment session by going through all questionnaires completed by the parent. The reasons why the parent did not answer all the questions will be discussed and collected, and the assessment and questionnaires at which the missing data occurred will be noted in the feasibility form.
Standard deviations of the main outcome to be evaluated in the full RCT | 2 weeks following the post-intervention wave of assessments (T1).
  The Variability score from the K-CPT2 is the main outcome of the future RCT. This data from the feasibility study will allow us to calculate the required standard deviation to be considered in the future RCT in accordance with the minimally clinical important difference (MCID) that should be measured between T0 and T1 for the yoga group.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Centre hospitalier universitaire Sainte-Justine, Montreal, Quebec
  - Centre universtaire de santé McGill, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marelli AJ, Ionescu-Ittu R, Mackie AS, Guo L, Dendukuri N, Kaouache M. Lifetime prevalence of congenital heart disease in the general population from 2000 to 2010. Circulation. 2014 Aug 26;130(9):749-56. doi: 10.1161/CIRCULATIONAHA.113.008396. Epub 2014 Jun 18. PMID 24944314
- [Background] Wang CC, Weng WC, Chang LY, Chang HY, Wu MH, Wang JK, Lu CW, Lin MT, Chen CA, Chiu SN. Increased prevalence of inattention-related symptoms in a large cohort of patients with congenital heart disease. Eur Child Adolesc Psychiatry. 2021 Apr;30(4):647-655. doi: 10.1007/s00787-020-01547-y. Epub 2020 May 11. PMID 32394091
- [Background] Lepage C, Gaudet I, Doussau A, Vinay MC, Gagner C, von Siebenthal Z, Poirier N, Simard MN, Paquette N, Gallagher A. The role of parenting stress in anxiety and sleep outcomes in toddlers with congenital heart disease. Front Pediatr. 2023 Jan 6;10:1055526. doi: 10.3389/fped.2022.1055526. eCollection 2022. PMID 36683797
- [Background] Gaudet I, Paquette N, Bernard C, Doussau A, Harvey J, Beaulieu-Genest L, Pinchefsky E, Trudeau N, Poirier N, Simard MN, Gallagher A; Clinique d'Investigation Neuro-Cardiaque (CINC) interdisciplinary team. Neurodevelopmental Outcome of Children with Congenital Heart Disease: A Cohort Study from Infancy to Preschool Age. J Pediatr. 2021 Dec;239:126-135.e5. doi: 10.1016/j.jpeds.2021.08.042. Epub 2021 Aug 27. PMID 34454950
- [Background] Lisanti AJ. Parental stress and resilience in CHD: a new frontier for health disparities research. Cardiol Young. 2018 Sep;28(9):1142-1150. doi: 10.1017/S1047951118000963. Epub 2018 Jul 11. PMID 29991369
- [Background] Mak CK, Whittingham K, Boyd RN. Experiences of children and parents in MiYoga, an embodied mindfulness yoga program for cerebral palsy: A mixed method study. Complement Ther Clin Pract. 2019 Feb;34:208-216. doi: 10.1016/j.ctcp.2018.12.006. Epub 2018 Dec 19. PMID 30712729
- [Background] Weaver LL, Darragh AR. Systematic Review of Yoga Interventions for Anxiety Reduction Among Children and Adolescents. Am J Occup Ther. 2015 Nov-Dec;69(6):6906180070p1-9. doi: 10.5014/ajot.2015.020115. PMID 26565100
- [Background] Cohen SCL, Harvey DJ, Shields RH, Shields GS, Rashedi RN, Tancredi DJ, Angkustsiri K, Hansen RL, Schweitzer JB. Effects of Yoga on Attention, Impulsivity, and Hyperactivity in Preschool-Aged Children with Attention-Deficit Hyperactivity Disorder Symptoms. J Dev Behav Pediatr. 2018 Apr;39(3):200-209. doi: 10.1097/DBP.0000000000000552. PMID 29538185
- [Derived] Simard MN, Lepage C, Gaudet I, Paquette N, Doussau A, Poirier NC, Beauchamp MH, Cote SM, Pinchefsky E, Brossard-Racine M, Masse B, Gallagher A. A Parent-child yoga intervention for reducing attention deficits in children with congenital heart disease: the Yoga for Little Hearts Feasibility Study Protocol. BMJ Open. 2023 Oct 17;13(10):e079407. doi: 10.1136/bmjopen-2023-079407. PMID 37848299